CLINICAL TRIAL: NCT07172763
Title: The Pressure Relieving Capacity of Siliconepads Compared to Felted Foam to Relieve Caput Metatarsal 2 in a Population With Diabetes at High Risk of Foot Ulcerations
Brief Title: The Pressure Relieving Capacity of Siliconepads Compared to Felted Foam to Relieve Caput Metatarsal 2 in a Population With Diabetes
Acronym: Siliconepads
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, DienstThoracaleEnVasculaireHeelkunde, Prof. Dr. Caren Randon, University Hospital, Ghent
Other Study IDs: ONZ-2024-0628
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diabete Mellitus; Peripheral Neuropathy
Keywords: Diabetes; Sensory peripheral neuropathy; Siliconepads; Felted foam; Plantar pressure measurement
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Siliconepad — Plantar pressure measurement
Device: Felted foam — Plantar pressure measurement

SUMMARY:
To evaluate the clinical effectiveness of siliconepads and if they could be an alternative to felted foam used in offloading high risk pressure areas in the plantar forefoot region using plantar pressure measurements.

Also user experience will be evaluated which is an important criterion in the use of this new type of offloading. Comfort, convenience and functionality of both felted foam and siliconepads will be tested to evaluate if siliconepads are more appropriate then felted foam.

DETAILED DESCRIPTION:
People with diabetes mellitus (DM) experience increased pressure under the plantar surface of the foot because of morphological, muscular and sensory abnormalities.

One third of these people have deformed feet, usually due to diabetic neuropathy, which causes localized increases in plantar pressure, particularly on the plantar side of the forefoot, where the risk of foot ulcers is high.

Custom-made therapeutic shoes and arch supports are recommended and are part of standard care for patients with foot deformities and a history of ulceration. The pressure under a human foot can be measured using a technique called Pedobarography or plantar pressure measurement, which uses insole- or platform-based pressure and force systems.

Pedobarographic measurements quantify the vertical load experienced by the foot when walking barefoot or with footwear by measuring the pressure on the plantar side. This makes it possible to identify any functional abnormalities in the structure and function of the dynamic foot. Wearing shoes with or without arch supports was reported to reduce peak pressure by 17 to 52% compared to walking barefoot. Furthermore, proof-of-principle studies have shown that reducing peak pressure on the plantar surface to less than 200 kPa (or by at least 25%) halves the risk of ulcer recurrence in people with diabetes over an 18-month period.

Felted foam therapy is, in addition to insoles and shoes, a complementary conservative treatment that facilitates this pressure relief. Felt consists of compressed wool in various thicknesses that distributes the increased pressure over a larger surface area, thereby reducing the peak pressure at a specific point. The location of the peak pressure is then relieved by the felt with a recess at this zone, whereby the pressure is distributed over the surface.

Felted foam, which has been the 3rd offloading method when it comes to local pressure relief after removable and non-removable knee-high devices, has many advantages but also its limitations. The material needs to be replaced weekly but in reality is often replaced every two days because the effect of the felt is limited in time. The thickness of the original felt decreases with wear and the material must not get wet.

Siliconepads, specifically designed for this study (Remedicare, Netherlands), with a CE certificate, could be more resistant than felt and a game changer in the offloading around the ulcer. These siliconepads are now used in treatment of skin tears and adapted for this study so this can be used and applied similarly to felted foam.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes, Peripheral neuropathy, able to walk 5 minutes, able to sign informed consent

Exclusion Criteria:

* No diabetes, No neuropathy, not able to walk without walking aid, not able to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with peripheral neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Plantar pressure reduction | 48 hours
  Achieve a plantar pressure decrease of 25%, leading to less than 200kpa under the 2nd caput metatarsal region after wearing siliconepads in comparison to barefoot plantar pressure measurement at baseline and after 48 hours.
  Achieve a plantar pressure decrease of 25% or less then 200kpa in the 2nd caput metatarsal region after wearing felted foam in comparison to barefoot plantar pressure measurement at baseline and after 48 hours.

IPD SHARING:
Plan to Share IPD: Undecided